CLINICAL TRIAL: NCT06051708
Title: Risk Factors And Outcomes Of Hospital Acquired Acute Kidney Injury: A Tertiary Health Care Center Experience
Brief Title: Risk Factors And Outcomes Of Hospital Acquired AKI
Status: Completed | Type: Observational
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mohamed Mamdouh Mahmoud Mohamed Elsayed , MD, Lecturer, Alexandria University
Other Study IDs: Hospiat Acq. AKI
Record Dates: First submitted 2023-09-17; First posted 2023-09-25 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: AKI - Acute Kidney Injury
Keywords: AKI; Hospital Acquired; risk factors; outcomes
MeSH Terms: conditions — Acute Kidney Injury | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AKI group: patients who are hospitalized and develop acute kidney injury after 48 hours from admission
  Interventions: Other: standard AKI care bundle
- no AKI group: patients who are hospitalized and do not develop acute kidney injury after 48 hours from admission till discharge
  Interventions: Other: standard care for hospitalized patients

INTERVENTIONS:
Other: standard AKI care bundle — AKI care bundle include use of iv fluids, diuretics, antihyperkalemic drugs, sodium bicarbonate, antibiotics in septic patients.
  Groups: AKI group
Other: standard care for hospitalized patients — this includes iv fluids, diuretics, antibiotics in septic patients, other measures according to original disease
  Groups: no AKI group

SUMMARY:
The aim of the study is to assess the common risk factors for development of hospital acquired acute kidney injury among hospitalized patients in Alexandria Main University hospital and their outcomes.

DETAILED DESCRIPTION:
Hospital-acquired AKI (HAAKI) is defined as acute renal insult occurring 48 hours or more after admission to a health care facility and It is estimated to occur in 13-18% of hospitalized patients. The early diagnosis of HAAKI reflects on improvement in morbidity and mortality rates especially in developing countries which goes parallel with the goal The International Society of Nephrology (ISN) to eliminate preventable or treatable deaths from AKI by 2025, the "0 by 25" initiative.

Data concerning the spectrum of acute kidney injury (AKI) in Egypt are generally scarce.

ELIGIBILITY:
Inclusion Criteria:

1. Fulfilment of definition of acute kidney injury according to KDIGO reference.
2. Age more than 18 years.

Exclusion Criteria:

1. Mentally or physically unfit patients.
2. Patients who developed acute kidney injury within 48 hours of admission to hospital.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This research is a prospective cohort study that will include hospitalized patients in Alexandria Main University Hospital (in non-intensive care unit sittings) admitted over a period of sixteen weeks.
  Patients will be divided into two groups:
  Group (A) : patients who are hospitalized and develop acute kidney injury after 48 hours from admission.
  Group (B) : patients who are hospitalized and do not develop acute kidney injury after 48 hours from admission till discharge.
  All participants will be followed till discharge and after 3 months to assess outcomes.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Recovery of kidney functions | 12 weeks
  (improvement of eGFR, serum creatinine to normal or previous baseline).

SECONDARY OUTCOMES:
progression to chronic kidney disease. | 12 weeks
  deterioration of kidney functions ( creatinine, eGFR)
mortality | 12 weeks
  death
Need for renal replacement therapy | 12 weeks
  different modalities of RRT

CONTACTS AND LOCATIONS:
Overall Officials: Hala S ElWakil, MD, Principal Investigator — professor; yasmine s naga, MD, Study Chair — ASS. prof; Mohamed mamdouh Elsayed, MD, Study Chair — Lecturer; sara R Nagib, MBBCh, Study Chair — Resident
Locations (1):
- Faculty of Medicine, Aexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Singh TB, Rathore SS, Choudhury TA, Shukla VK, Singh DK, Prakash J. Hospital-acquired acute kidney injury in medical, surgical, and intensive care unit: A comparative study. Indian J Nephrol. 2013 Jan;23(1):24-9. doi: 10.4103/0971-4065.107192. PMID 23580801
- [Background] Sawhney S, Mitchell M, Marks A, Fluck N, Black C. Long-term prognosis after acute kidney injury (AKI): what is the role of baseline kidney function and recovery? A systematic review. BMJ Open. 2015 Jan 6;5(1):e006497. doi: 10.1136/bmjopen-2014-006497. PMID 25564144
- [Background] Hsu CN, Lee CT, Su CH, Wang YL, Chen HL, Chuang JH, Tain YL. Incidence, Outcomes, and Risk Factors of Community-Acquired and Hospital-Acquired Acute Kidney Injury: A Retrospective Cohort Study. Medicine (Baltimore). 2016 May;95(19):e3674. doi: 10.1097/MD.0000000000003674. PMID 27175701
- [Background] Ponce D, Balbi A. Acute kidney injury: risk factors and management challenges in developing countries. Int J Nephrol Renovasc Dis. 2016 Aug 22;9:193-200. doi: 10.2147/IJNRD.S104209. eCollection 2016. PMID 27578995